CLINICAL TRIAL: NCT02697214
Title: Accuracy of Commercially Available Heart Rate Monitors: A Prospective Study
Brief Title: Accuracy of Commercially Available Heart Rate Monitors
Acronym: HRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Marc Gillinov, MD, MD, The Cleveland Clinic
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 15-718
Record Dates: First submitted 2016-02-24; First posted 2016-03-03 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: commercial heart rate monitors; accuracy; ECG; varying degrees of exertion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Apple Watch (Active Comparator): Apple Watch heart rate monitoring device worn with standard ECG, Polar H7 chest monitor and one other wrist monitoring device .
  Interventions: Device: Apple Watch
- Fitbit Charge HR (Active Comparator): Fitbit Charge HR heart rate monitoring device worn with standard ECG, Polar H7 chest monitor and one other wrist monitoring device.
  Interventions: Device: Fitbit Charge HR
- Mio Fuse (Active Comparator): Mio Fuse heart rate monitoring device worn with standard ECG, Polar H7 chest monitor and one other wrist monitoring device.
  Interventions: Device: Mio Fuse
- Basis Peak (Active Comparator): Basis Peak heart rate monitoring device worn with standard ECG, Polar H7 chest monitor and one other wrist monitoring device.
  Interventions: Device: Basis Peak

INTERVENTIONS:
Device: Fitbit Charge HR — Fitbit Charge HR heart rate monitoring device compared to ECG and Polar H7
  Arms: Fitbit Charge HR
Device: Apple Watch — Apple Watch heart rate monitoring device compared to ECG and Polar H7
  Arms: Apple Watch
Device: Mio Fuse — Mio Fuse heart rate monitoring device compared to ECG and Polar H7
  Arms: Mio Fuse
Device: Basis Peak — Basis Peak heart rate monitoring device compared to ECG and Polar H7
  Arms: Basis Peak

SUMMARY:
Over the last two decades, there has been a proliferation of commercially available heart rate monitors. Recognizing that elite athletes often use heart rate to monitor training and assess aerobic fitness, fitness companies have offered a variety of heart rate monitoring systems to the general public. Recently, there has been a move from monitors that rely on chest straps to measure electrical activity toward more convenient, wrist-worn monitors that employ optical sensing technology similar to that used for pulse oximetry. While the accuracy of chest strap monitors has been assessed in a variety of studies, there is no data concerning the accuracy of wrist-worn heart rate monitors. Assessment of the monitors' accuracy is important both for the subjects who rely upon these monitors to guide their athletic activity and for the physicians to whom these individuals report their heart rate readings.

DETAILED DESCRIPTION:
Physicians have long-used heart rate as an index of aerobic fitness and cardiovascular health. Resting heart rate has been linked to longevity and freedom from cardiovascular morbidity, and heart rate during exercise serves as a measure of aerobic capacity. In addition, heart rate recovery after exercise carries implications for an individuals' health.

Like physicians, coaches and athletic trainers employ heart rate measurement on a daily basis. In the athletic setting, heart rate during exercise is used as an indication of aerobic exertion. Elite athletes and their coaches often design workouts based upon achieved and targeted heart rates.

Once the province of physicians and elite athletes, heart rate monitoring has become widespread among the general public. In the nineteen eighties, fitness companies added heart rate monitors to their product lines. Systems employing a chest strap to monitor electrical activity, telemetry and a wrist-borne receiver became popular, and several controlled, scientific studies confirmed their accuracy.

More recently, manufacturers have marketed a new class of heart rate monitors that consist solely of wristwatch-style devices. These heart rate monitors use optical sensing technology to measure heart rate. While they offer convenience, their accuracy, particularly during exercise, is uncertain. A recent article in USA Today suggests that these wrist-worn monitors fail to provide accurate readings during exercise; however, to date there has been no rigorous scientific inquiry addressing this question.

The purpose of this study is to assess the accuracy of four popular, commercially available wrist-worn heart rate monitors under conditions of varying physical exertion.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Able and willing to exercise (walk/jog) for a total of fifteen minutes

Exclusion Criteria:

* Health issues that preclude or contraindicate walking and/or jogging, including cardiovascular, orthopedic, pulmonary and other conditions
* Presence of a cardiac pacemaker
* Known cardiovascular disease
* Known heart rhythm disorders
* Use of Beta-blockers or antiarrhythmic medications
* Tattoos around the wrist area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Gillinov, MD, Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 50 subjects wore 4 monitors each. i.e. EKG, H7 polar monitor, and 2 other randomly assigned heart rate monitors.
Units Other Than Participants: Heart Rate monitors
Groups:
- Apple Watch: Participants wore Polar H7 chest monitor, standard ECG and Apple Watch and one other wrist monitor.
- Fitbit Charge HR: Participants wore Polar H7 chest monitor, standard ECG and Fitbit Charge HR and one other wrist monitor.
- Mio Fuse: Participants wore Polar H7 chest monitor, standard ECG and Mio Fuse and one other wrist monitor.
- Basis Peak: Participants wore Polar H7 chest monitor and Basis Peak and one other wrist monitor.
- Polar HR: All participants wore Polar HR chest monitor
- Standard ECG: All participants wore standard ECG
Period: Overall Study
Arm/Group | Apple Watch | Fitbit Charge HR | Mio Fuse | Basis Peak | Polar HR | Standard ECG
Started (Each subject wore standard EKG, Polar H7 and 2 wrist monitoring devices) | 26; 26 Heart Rate monitors | 25; 25 Heart Rate monitors | 25; 25 Heart Rate monitors | 24; 24 Heart Rate monitors | 50; 50 Heart Rate monitors | 50; 50 Heart Rate monitors
Heart Rate at 2mph | 26; 26 Heart Rate monitors | 25; 25 Heart Rate monitors | 25; 25 Heart Rate monitors | 24; 24 Heart Rate monitors | 50; 50 Heart Rate monitors | 50; 50 Heart Rate monitors
Heart Rate at 3mph | 26; 26 Heart Rate monitors | 25; 25 Heart Rate monitors | 25; 25 Heart Rate monitors | 24; 24 Heart Rate monitors | 50; 50 Heart Rate monitors | 50; 50 Heart Rate monitors
Heart Rate at 4mph | 26; 26 Heart Rate monitors | 25; 25 Heart Rate monitors | 25; 25 Heart Rate monitors | 24; 24 Heart Rate monitors | 50; 50 Heart Rate monitors | 50; 50 Heart Rate monitors
Heart Rate at 6mph | 26; 26 Heart Rate monitors | 25; 25 Heart Rate monitors | 25; 25 Heart Rate monitors | 24; 24 Heart Rate monitors | 50; 50 Heart Rate monitors | 50; 50 Heart Rate monitors
Completed | 26; 26 Heart Rate monitors | 25; 25 Heart Rate monitors | 25; 25 Heart Rate monitors | 24; 24 Heart Rate monitors | 50; 50 Heart Rate monitors | 50; 50 Heart Rate monitors
Not Completed | 0; 0 Heart Rate monitors | 0; 0 Heart Rate monitors | 0; 0 Heart Rate monitors | 0; 0 Heart Rate monitors | 0; 0 Heart Rate monitors | 0; 0 Heart Rate monitors

BASELINE CHARACTERISTICS:
Population: Analysis was done per device. Each participant (50 total) wore 2 wrist devices in addition to a Polar H7 chest monitor and standard ECG monitor. Accuracy of the wrist devices was assessed using Concordance Correlation Coefficient.
Units Other Than Participants: Heart Rate Monitors
Groups:
- Apple Watch: Apple Watch heart rate monitoring device.
  Apple Watch: Apple Watch heart rate monitoring device.
- Fitbit Charge HR: Fitbit Charge HR heart rate monitoring device.
  Fitbit Charge HR: Fitbit Charge HR heart rate monitoring device.
- Mio Fuse: Mio Fuse heart rate monitoring device.
  Mio Fuse: Mio Fuse heart rate monitoring device.
- Basis Peak: Basis Peak heart rate monitoring device.
  Basis Peak: Basis Peak heart rate monitoring device.
- Total: Total of all reporting groups
Arm/Group | Apple Watch | Fitbit Charge HR | Mio Fuse | Basis Peak | Total
Number analyzed (Participants) | 26 | 25 | 25 | 24 | 50
Number analyzed (Heart Rate Monitors) | 26 | 25 | 25 | 24 | 100
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 25 | 25 | 24 | 50
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Female | 19 | 12 | 14 | 13 | 29
  Male | 7 | 13 | 11 | 11 | 21
Region of Enrollment [Number; unit: participants] — Population: As each participant was assigned to wear two wrist-worn heart rate monitors.
  participants
    United States | 26 | 25 | 25 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Measuring the Accuracy of Commercial Heart Rate Monitors.
Description: The purpose of this study is to assess the accuracy of four popular, commercially available wrist-worn heart rate monitors compared to the current gold standard of a ECG using Lin's Concordance Correlation Coefficient.
Time Frame: 20 minutes
Population: All participants are represented in the analysis population.
Measure: Number (95% Confidence Interval); unit: Correlation Coefficient
Units Other Than Participants: Heart Rate Monitors
Arm/Group | Apple Watch | Fitbit Charge HR | Mio Fuse | Basis Peak
Number analyzed (Participants) | 26 | 25 | 25 | 24
Number analyzed (Heart Rate Monitors) | 26 | 25 | 25 | 24
Correlation Coefficient | .91 [.884 to .929] | .84 [.791 to .872] | .91 [.882 to .929] | .83 [.779 to .865]

ADVERSE EVENTS:
Time Frame: 1 day. Adverse events were collected during the active portion of the trial which constituted the time on the treadmill.
Arm/Group | Apple Watch | Fitbit Charge HR | Mio Fuse | Basis Peak
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25 | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/25 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes